CLINICAL TRIAL: NCT07038135
Title: Formulation, Phytochemical Characterization, and Clinical Assessment of a Novel Natural Supplement Targeting Body Composition in Physically Active Individuals: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Formulation, Phytochemical Characterization, and Clinical Assessment of a Novel Natural Supplement Targeting Body Composition in Physically Active Individuals
Acronym: NSCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sulaimany Polytechnic university (Other)
Responsible Party: Principal Investigator, Farhang Hameed Awlqadr, Researcher, Sulaimany Polytechnic university
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPU2025NUTR01
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Improving Body Composition; Novel Natural Gym Nutrient Formulation; Increase Muscle Mass; Reduce Body Fat Percentage; Enhancing Metabolic Health and Athletic Performance
Keywords: Body composition; Muscle mass; Natural supplement; Herbal formulation; Randomized controlled trial; Placebo-controlled trial; Antioxidant capacity

STUDY DESIGN:
Intervention Model Description: This is a parallel study design, where participants are randomly assigned to one of two groups: the treatment group receiving the natural supplement (NNS) and the control group receiving a placebo. Both groups are followed concurrently for the duration of the 8-week study period to assess the intervention's impact on body composition, including muscle mass and fat percentage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind, placebo-controlled study, the following parties are masked:
  Participants: They are unaware of whether they are receiving the Novel Natural Supplement (NNS) or the placebo, ensuring unbiased reporting of results.
  Care Providers: The individuals administering the treatment or placebo are blinded to prevent any bias in delivering the intervention.
  Investigators: The researchers responsible for data collection and analysis do not know which participants are in the treatment or placebo groups, reducing bias in assessments and interpretation.
  Outcomes Assessors: Those measuring body composition and other health parameters are blinded to participant group assignments to ensure unbiased measurement and analysis.
  This rigorous blinding process helps ensure that the outcomes are not influenced by expectations or biases from any party involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Natural Supplement (NNS) Group (Experimental): Participants in this arm received a daily 30-gram dose of the Novel Natural Supplement (NNS), a multi-ingredient formula containing whey protein, pea protein, oats, sweet potato, flaxseed, chia seeds, spinach powder, cardamom, green tea extract, beetroot powder, and stevia. The intervention lasted for 8 weeks to assess its effect on body composition and metabolic health.
  Interventions: Dietary Supplement: Novel Natural Supplement (NNS); Dietary Supplement: Placebo
- Placebo Group (Placebo Comparator): Participants in this arm received a daily 30-gram dose of a placebo consisting of maltodextrin, microcrystalline cellulose, and beetroot powder, matched in appearance, flavor, and texture to the NNS. The intervention lasted for 8 weeks to serve as a control for the trial.
  Interventions: Dietary Supplement: Novel Natural Supplement (NNS); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Novel Natural Supplement (NNS) — Multi-ingredient formula including whey protein, pea protein, oats, sweet potato, flaxseed, chia seeds, spinach powder, cardamom, green tea extract, beetroot powder, and stevia. Administered daily for 8 weeks.
  Other Names: Experimental
Dietary Supplement: Placebo — A placebo containing maltodextrin, microcrystalline cellulose, and beetroot powder, matched in appearance, flavor, and texture to the NNS. Administered daily for 8 weeks.

SUMMARY:
This study aims to evaluate the efficacy of a novel natural gym nutrient formulation (NNS) in improving body composition in physically active individuals. The formulation consists of a multi-ingredient blend of natural ingredients including whey protein, pea protein, oats, sweet potato, flaxseed, chia seeds, spinach powder, green tea extract, and beetroot powder. These ingredients are carefully selected for their potential to enhance muscle mass, reduce body fat, and improve metabolic health.

The study follows a randomized, double-blind, placebo-controlled design where participants are randomly assigned to receive either the NNS or a placebo (PLA). Both the NNS and PLA are identical in appearance to maintain the blinding of both the participants and the investigators. The trial is conducted over 8 weeks, with daily supplementation and body composition assessments (muscle mass, fat percentage, body water content) being conducted at baseline and at the end of the intervention. The study also includes analysis of the formulation's chemical properties, antioxidant capacity, and bioactive compounds to validate its effectiveness.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial assessed the efficacy of a novel, multi-ingredient natural supplement (NNS) designed to improve body composition and metabolic health in endurance-trained individuals. The NNS formulation combines plant-based proteins, dietary fibers, polyphenols, and antioxidant-rich botanicals with the aim of enhancing lean mass, reducing body fat, and supporting cardiopulmonary function. The active ingredients include whey protein, pea protein, oats, sweet potato, flaxseed, chia seeds, spinach powder, cardamom, green tea extract, beetroot powder, and stevia.

Prior to clinical assessment, the formulation underwent detailed chemical characterization, including analysis of physicochemical properties (pH, acidity, °Brix), proximate composition (fat and protein content), mineral profile (via ICP-OES), fatty acid composition (via GC-FID), antioxidant capacity (DPPH and ABTS assays), and bioactive compound identification (GC-MS). The formulation demonstrated high protein content, a favorable fatty acid profile rich in omega-3s, potent antioxidant activity, and the presence of bioactive compounds with anti-inflammatory and muscle-supportive properties.

In the clinical phase, participants were randomly assigned to consume either the NNS or a placebo (matched in appearance, flavor, and texture) daily for 8 weeks. Blinding was maintained for participants, care providers, investigators, and outcome assessors. Body composition was assessed via bioelectrical impedance analysis, alongside measurements of oxygen saturation, heart rate, and serum metabolic markers. The study aimed to provide scientific validation for the role of natural, protein-rich, multi-ingredient supplements in promoting muscle accretion, reducing body weight and BMI, improving metabolic markers, and supporting cardiopulmonary health in physically active individuals

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 45 years
* Body Mass Index (BMI) between 18.5 and 29.5 kg/m²
* Engaging in endurance training at least 3 times per week
* Ability to provide written informed consent prior to participation

Exclusion Criteria:

* Current smoker
* Use of assistive walking devices
* Chronic use of analgesic or anti-inflammatory medications
* Diagnosed with any of the following conditions:
* - Diabetes mellitus
* - Cardiovascular disease (including recent myocardial infarction or hypertension requiring more than two medications)
* - Congestive heart failure
* - Renal disease
* - Previous stroke
* Active musculoskeletal injury and/or severe osteoarthritis
* Significant weight change (more than ±4 kg) in the 8 weeks prior to the study
* Unable or unwilling to comply with study requirements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass (kg or %) | 8 weeks (post-intervention)
  The primary objective of this study is to evaluate the effect of the Novel Natural Supplement (NNS) on muscle mass in physically active individuals. Muscle mass will be assessed using bioelectrical impedance analysis (BIA) at baseline and at the end of the 8-week intervention period.

SECONDARY OUTCOMES:
Change in body fat percentage (%) | 8 weeks (post-intervention)
  The secondary outcome is to assess the effect of NNS on body fat percentage. Body fat will be measured using bioelectrical impedance analysis (BIA) at baseline and after 8 weeks of supplementation.
Change in Body Mass Index (BMI) (kg/m²) | 8 weeks (post-intervention)
  BMI will be calculated using participants' weight and height at baseline and after 8 weeks of supplementation. This measure will help assess changes in body composition (i.e., weight and fat mass) relative to height and can provide additional insights into the overall effect of the intervention on participants' physical health.

OTHER OUTCOMES:
Change in weight (kg) | 8 weeks (post-intervention)
  he effect of the Novel Natural Supplement (NNS) on body weight will be assessed by measuring the participants' weight at baseline and after 8 weeks of supplementation. This outcome will help evaluate whether the supplement contributes to weight loss or gain, depending on changes in muscle mass and fat percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Halabja Technical college, Sulaymaniyah, Halabja Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) to be shared will include de-identified data on body composition (muscle mass, fat percentage, body water content), weight, BMI, and blood glucose levels from participants who have completed the 8-week study. The data will be shared in a secure, anonymized format and will only be available to qualified researchers after study completion. Access will be granted through a formal data request process, ensuring privacy and compliance with ethical standards. All data will be stored and shared through a secure data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The individual participant data (IPD) and supporting information (such as study protocol, statistical analysis plan, informed consent form, and clinical study report) will be made available 6 months after the completion of data collection, ensuring all study results are finalized and analyzed. The data will remain accessible for a period of 5 years from the date of publication or final analysis to allow for secondary analyses by qualified researchers.
Access Criteria: The IPD and supporting information will be accessible to qualified researchers affiliated with academic institutions or research organizations, provided they submit a formal data request. Access will be granted to de-identified data related to body composition, weight, BMI, and other clinical measures as outlined in the study protocol. Researchers will be able to access the data via a secure data-sharing platform, and access will be granted only after ethical approval or a data-sharing agreement is in place to ensure compliance with privacy regulations.

REFERENCES:
- [Background] Nehmi-Filho V, Santamarina AB, de Freitas JA, Trarbach EB, de Oliveira DR, Palace-Berl F, de Souza E, de Miranda DA, Escamilla-Garcia A, Otoch JP, Pessoa AFM. Novel nutraceutical supplements with yeast beta-glucan, prebiotics, minerals, and Silybum marianum (silymarin) ameliorate obesity-related metabolic and clinical parameters: A double-blind randomized trial. Front Endocrinol (Lausanne). 2023 Jan 27;13:1089938. doi: 10.3389/fendo.2022.1089938. eCollection 2022. PMID 36778595
- [Background] Nederveen JP, Mastrolonardo AJ, Xhuti D, Di Carlo A, Manta K, Fuda MR, Tarnopolsky MA. Novel Multi-Ingredient Supplement Facilitates Weight Loss and Improves Body Composition in Overweight and Obese Individuals: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Nutrients. 2023 Aug 23;15(17):3693. doi: 10.3390/nu15173693. PMID 37686725